CLINICAL TRIAL: NCT05563220
Title: A Phase 1b/2, Open-Label Umbrella Study To Evaluate Safety And Efficacy Of Elacestrant In Various Combination In Patients With Metastatic Breast Cancer
Brief Title: Open-Label Umbrella Study To Evaluate Safety And Efficacy Of Elacestrant In Various Combination In Participants With Metastatic Breast Cancer
Acronym: ELEVATE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STML-ELA-0222
Record Dates: First submitted 2022-09-22; First posted 2022-10-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; Alpelisib; Everolimus; ribociclib; palbociclib; capivasertib; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1b Arm A: elacestrant with alpelisib (Experimental): Elacestrant Dihydrochloride 300 milligrams (mg) or 400 mg + Alpelisib 150 mg to 250 mg
  Interventions: Drug: Elacestrant; Drug: Alpelisib
- Phase 1b Arm B: elacestrant with everolimus (Experimental): Elacestrant Dihydrochloride 300 mg or 400 mg + Everolimus 5.0 mg, 7.5 mg or possibly 10 mg
  Interventions: Drug: Elacestrant; Drug: Everolimus
- Phase 1b Arm C: elacestrant with abemaciclib or ribociclib: (Experimental): Elacestrant Dihydrochloride 100 mg, 200 mg, 300 mg + Ribociclib 400 mg or possibly 600 mg
  The RP2D for the combination of elacestrant and abemaciclib is evaluated in the ongoing ELECTRA trial (ClinicalTrials.gov Identifier: NCT04791384)
  Interventions: Drug: Elacestrant; Drug: Ribociclib; Drug: Abemaciclib
- Phase 1b Arm D: elacestrant with either palbociclib, abemaciclib, or ribociclib (no prior CDK4/6i) (Experimental): Elacestrant Dihydrochloride 300 mg or 400 mg + Palbociclib 100 mg,125 mg or the RP2D for the combination of elacestrant and abemaciclib is evaluated in the ongoing ELECTRA trial (ClinicalTrials.gov Identifier: NCT04791384)
  Elacestrant 86 mg, 172 mg, 258 mg + Ribociclib 400 mg or possibly 600 mg
  Interventions: Drug: Elacestrant; Drug: Ribociclib; Drug: Palbociclib; Drug: Abemaciclib
- Phase 1b Arm E: (Experimental): Elacestrant Dihydrochloride 300 mg, 400 mg + Capivasertib 200 mg, 320 mg, 400 mg
  Interventions: Drug: Elacestrant; Drug: Capivasertib

INTERVENTIONS:
Drug: Elacestrant — Elacestrant 86 mg, 172 mg, 258 mg or 345 mg once daily in cycles of 28 days
Drug: Alpelisib — Alpelisib 150 mg or 250 mg once daily in cycles of 28 days
  Other Names: Piqray
  Arms: Phase 1b Arm A: elacestrant with alpelisib
Drug: Everolimus — Everolimus 5 mg, 7.5 mg, or 10 mg once daily in cycles of 28 days
  Other Names: Afinitor
  Arms: Phase 1b Arm B: elacestrant with everolimus
Drug: Ribociclib — Ribociclib 400 mg or 600 mg once daily for 21 days followed by 7 days off in cycles of 28 days
  Other Names: Kisqali
  Arms: Phase 1b Arm C: elacestrant with abemaciclib or ribociclib:; Phase 1b Arm D: elacestrant with either palbociclib, abemaciclib, or ribociclib (no prior CDK4/6i)
Drug: Palbociclib — Palbociclib 100 mg or 125 mg once daily for 21 days followed by 7 days off in cycles of 28 days
  Other Names: Ibrance
  Arms: Phase 1b Arm D: elacestrant with either palbociclib, abemaciclib, or ribociclib (no prior CDK4/6i)
Drug: Capivasertib — Capivasertib 200 mg or 320 mg or 400 mg twice daily for 4 days on, 3 days off in cycles of 28 days
  Other Names: Truqap
  Arms: Phase 1b Arm E:
Drug: Abemaciclib — Abemaciclib 100 mg or 150 mg twice daily in cycles of 28 consecutive days
  Other Names: Verzenio
  Arms: Phase 1b Arm C: elacestrant with abemaciclib or ribociclib:; Phase 1b Arm D: elacestrant with either palbociclib, abemaciclib, or ribociclib (no prior CDK4/6i)

SUMMARY:
This is a multicenter, Phase 1b/2 trial in participants with estrogen receptor positive/human epidermal growth factor receptor 2 negative (ER+/HER2-) advanced/metastatic breast cancer. The phase 1b part of the trial will determine the recommended Phase 2 dose (RP2D) of elacestrant when administered in combination with alpelisib, everolimus, palbociclib, capivasertib, and ribociclib. The Phase 2 part of the trial will evaluate the efficacy and safety of the various combinations.

DETAILED DESCRIPTION:
This is a multicenter, Phase 1b/2 trial. The Phase 1b aims at selecting the RP2D dose, defined as a dose that is associated with less than 33% of participants experiencing a dose-limiting toxicity (DLT) of elacestrant when administered in combination with alpelisib, everolimus, palbociclib, ribociclib, and capivasertib that is, ≤1 participant experiencing a DLT out of 6 DLT-evaluable participants. For each combination, this phase will have approximately 3 cohorts of up to 6 DLT-evaluable participants each. The total number of DLT-evaluable participants in all the combinations will be up to 125.

The Phase 2 part of the trial will evaluate the efficacy and safety of the various combinations.

The treatment arms will be:

* Arm A: 50 participants: elacestrant with alpelisib;
* Arm B: 50 participants: elacestrant with everolimus;
* Arm C: 60 participants (30 participants in each combination): elacestrant with either abemaciclib or ribociclib;
* Arm D: 90 participants (30 participants in each combination): elacestrant with either palbociclib, abemaciclib, or ribociclib;
* Arm E: 60 participants: elacestrant with capivasertib

Phase 1b will have a total of 125 participants, while Phase 2 will have 310 participants for all treatment arm combinations.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has signed the informed consent before all study specific activities are conducted.
2. Women or men aged ≥18 years (or the minimum age of consent in accordance with the local law), at the time of informed consent signature. Female participants may be of any menopausal status.

   * Postmenopausal status is defined as follows or in accordance with local regulations:

     1. Age ≥60 years or
     2. Age <60 years and amenorrhea for 12 or more months (without an alternative cause) and follicle-stimulating hormone value and an estradiol level within the postmenopausal range per local laboratory reference or
     3. Documentation of bilateral oophorectomy, at least 1 month before first dose of trial therapy.
   * Premenopausal and perimenopausal women (who do not fit postmenopausal criteria) and men must be receiving a luteinizing hormone-releasing hormone (LHRH) agonist and must be initiated at least 3 weeks (4 depending on local label) before the start of trial therapy and are planning to continue LHRH agonist treatment during the study treatment.
3. Histopathological or cytological confirmed ER+, HER2-, breast cancer, per local laboratory, as per the American Society of Clinical Oncology/College of American Pathologists guidelines. Note: In the context of this trial, ER status will be considered positive if ≥10% of tumor cells demonstrate positive nuclear staining by immunohistochemistry, with or without progesterone positivity.
4. Documented radiological disease progression during or after the most recent therapy.
5. At least 1 measurable lesion as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Tumor lesions previously irradiated or subjected to any locoregional treatment will only be considered measurable if there is clear, documented progression at the treated site. For participants with bone only disease, lesions: must be lytic or mixed (lytic + blastic / sclerotic), confirmed and accurately assessed by computed tomography or magnetic resonance imaging, and must have an identifiable soft tissue component meeting the definition of measurability per RECIST v1.1. Note: participants with blastic / sclerotic bone lesions only are not eligible.
6. Eastern Cooperative Oncology Group performance status of 0 or 1.
7. Participant has adequate bone marrow and organ function, as defined by the following laboratory values:

   1. Absolute neutrophil count ≥1.5 × 10^9/liter (L)
   2. Platelets ≥100 × 10^9/L
   3. Hemoglobin ≥9.0 grams/deciliter (g/dL)
   4. Creatinine is ≤ 1.5 x upper limit of normal (ULN) or if creatinine is > 1.5 x ULN, then creatinine clearance must be ≥50 milliliters/minute based on the Cockcroft-Gault formula. Note: C-G formula:

      * Creatinine clearance (male) = ([140-age in years] × weight in kilograms [kg])/ ([serum creatinine in milligrams/deciliter (mg/dL)] × 72)
      * Creatinine clearance (female) = (0.85 × [140-age in years] × weight in kg)/ ([serum creatinine in mg/dL] × 72)

   f. Serum albumin ≥3.0 g/dL (≥30 g/L)

   g. In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN. If the participant has liver metastases, ALT and AST ≤ 5 × ULN

   h. Total serum bilirubin <1.5 × ULN except for participants with Gilbert's syndrome who may be included if the total serum bilirubin is ≤3.0 × ULN or direct bilirubin ≤ 1.5 × ULN.

Additional Criteria for the Alpelisib Combination (Phase 1b and Arm A): In general, the prescription information of the respective combination drug should be consulted for instructions/restrictions with respect to interactions with concomitant medications.

1. Phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) mutation by local laboratory assessment.
2. One or up to two prior hormonal therapies in the advanced or metastatic setting, one of which was in combination with a cyclin-dependent kinase targeting enzymes CDK4 and CDK6 (CDK4/6) inhibitor.

Additional Criteria for the Everolimus Combination (Phase 1b and Arm B), the Abemaciclib Combination (Arm C), the Ribociclib Combination (Phase 1b and Arm C), and the Palbociclib Combination (Phase 1b): One or up to two prior hormonal therapies in the advanced or metastatic setting, one of which was in combination with a CDK4/6 inhibitor.

Additional Criteria for the Palbociclib Combination (Arm D), the Abemaciclib Combination (Arm D), and the Ribociclib Combination (Arm D): One or up to two prior hormonal therapies in the advanced or metastatic setting.

Additional Criteria for Capivasertib Combination (Phase 1b and Arm E): Recruitment in this combination will occur only in countries where capivasertib is locally approved and available.

1. PIK3CA/AKT1/PTEN-alteration as detected by an FDA and/or locally approved test (local result).
2. One or up to two prior hormonal therapies in the advanced or metastatic setting or participants who have radiological evidence of breast cancer recurrence or progression within 12 months from the end of adjuvant treatment with endocrine therapy, as these participants are considered as first line relapsed participants. Prior CDK4/6i treatment is allowed but not required.

Exclusion Criteria:

1. Active or newly diagnosed central nervous system metastases, or meningeal carcinomatosis. Note: Participants with stable brain or subdural metastases are allowed if the participant has completed local therapy and was on a stable or decreasing dose of corticosteroids at baseline for management of brain metastasis for at least 4 weeks before starting treatment in this study. The dose must be ≤2.0 mg/day of dexamethasone or equivalent. Any signs (for example, radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
2. Participants with advanced, symptomatic visceral spread, who are at risk of life-threatening complications in the short term, including massive uncontrolled effusions (peritoneal, pleural, pericardial), pulmonary lymphangitis, or liver involvement >50%.
3. Prior chemotherapy or elacestrant in the advanced/metastatic setting.
4. Participants with known germline BRCA mutation without prior treatment with a PARP inhibitor before study entry.
5. Prior therapy with elacestrant or other investigational selective estrogen receptor degraders, or investigational alike agents such as selective estrogen receptor modulators, selective estrogen receptor covalent antagonists, complete estrogen receptor antagonists, and proteolysis-targeting chimeras, in the metastatic setting. Prior treatment with fulvestrant is not exclusionary, except for Arm E, as it is an approved medication.
6. Participant has a concurrent malignancy or history of invasive malignancy within 3 years of enrollment, except basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix that has completed curative therapy. Other malignancies with low risk of recurrence may be considered eligible with Sponsor approval.
7. Uncontrolled significant active infections.

   * Participants with hepatitis B virus and/or hepatitis C virus infection must have undetectable viral load during screening.
   * Participants known to be human immunodeficiency virus+ are allowed if they have undetectable viral load at baseline.
8. Documented pneumonitis/interstitial lung disease prior to Cycle 1 Day 1.
9. Major surgery within 28 days before starting trial therapy.
10. Inability to take oral medications, refractory or chronic nausea, gastrointestinal conditions (including significant gastric or bowel resection), history of malabsorption syndrome, or any other uncontrolled gastrointestinal condition that impact the absorption of the study drug.
11. Known intolerance to elacestrant or any of its excipients.
12. Pregnant and breast-feeding women are excluded from the study. In addition, women of childbearing potential are excluded who:

    * Within 28 days before starting trial therapy, did not use a highly effective method of contraception.
    * Do not agree to use a highly effective method of contraception (Appendix F) or abstain from heterosexual intercourse throughout the entire study period and for 120 days after trial therapy discontinuation.
13. Men or women who do not agree to abstain from donating sperm or ova, or to use a highly effective method of contraception, 28 days prior, during the course of the treatment period and for 120 days after the last dose of study treatment.
14. Participant is currently receiving or received any of the following medications prior to first dose of trial therapy:

    • Anti-cancer therapy within 14 days (28 days for anticancer antibody based treatment) or 5 half-lives, whichever is shorter.

    Please note: Toxicity from prior therapy must be resolved to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 Grade ≤1, except alopecia and peripheral sensory neuropathy (Grade ≤2).
    * Known strong or moderate inducers or inhibitors of cytochrome P450 (CYP) 3A4 within 14 days or 5 half-lives, whichever is shorter, (refer to https://drug-interactions.medicine.iu.edu/maintable.aspx or https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers).
    * Herbal preparations/medications within 7 days. These include, but are not limited to, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng.
    * Vaccination, including but not limited to vaccination against COVID-19, during the 7 days prior to starting trial therapy.
15. Evidence of ongoing alcohol or drug abuse as assessed by the investigator.
16. Any severe medical or psychiatric condition that, in the Investigator's opinion, would preclude the participant's participation in a clinical study.

Additional Criteria for the Alpelisib Combination (Phase 1b and Arm A):

1. Prior therapy with alpelisib or any other phosphoinositide 3-kinase (PI3K) inhibitor.
2. Type 1 diabetes or uncontrolled type 2 diabetes (fasting plasma glucose level of >140 mg/dL [7.7 millimole (mmol)/L], or glycosylated hemoglobin [HbA1c] level of >6.4%).
3. Known intolerance to alpelisib or any of its excipients.
4. Participant is currently receiving or received drugs known to be a breast cancer resistant protein inhibitor (for example, curcumin, cyclosporine A, eltrombopag, febuxostat, fostamatinib, rolapitant, teriflunomide) within 14 days or 5 half-lives, whichever is shorter, prior to first dose of trial therapy (refer to Table 5.2 of https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers).
5. Participant has ongoing osteonecrosis of the jaw from previous or concurrent treatment with bisphosphonates or denosumab

Additional Criteria for the Everolimus Combination (Phase 1b and Arm B):

1. Prior therapy with everolimus.
2. Known intolerance to everolimus or any of its excipients.

Additional Criteria for the Abemaciclib Combination (Arm C):

1. Prior therapy with abemaciclib in the advanced or metastatic setting. Adjuvant therapy with abemaciclib is also exclusionary.
2. Known intolerance to abemaciclib or any of its excipients.
3. History of deep vein thrombosis or pulmonary embolism (unless on anticoagulation), cerebrovascular accident, or myocardial infarction, in the past 6 months. Participants on anticoagulation should have been on a stable dose for at least 3 months prior to enrollment.

Additional Criteria for the Ribociclib Combination (Phase 1b and Arm C):

1. Prior therapy with ribociclib in the advanced or metastatic setting. Prior adjuvant therapy with ribociclib is also exclusionary.
2. Known intolerance to ribociclib or any of its excipients.
3. QTcF interval corrected by Fridericia formula (QTcF) values ≥450 milliseconds (msec).
4. Participants who already have or who are at significant risk of developing QTc prolongation, including participants with:

   * Long QT syndrome
   * Uncontrolled or significant cardiac disease including recent (6 months) myocardial infarction, congestive heart failure, unstable angina, and brady-arrhythmias
   * Electrolyte abnormalities (K+, Ca++, Phos, Mg++) ≥Grade 1
5. Participant is currently receiving or received drugs known to prolong QT interval within 14 days or 5 half-lives, whichever is shorter, before the first dose of trial therapy.

Additional Criteria for the Palbociclib Combination (Phase 1b):

1. Prior therapy with palbociclib in the advanced or metastatic setting.
2. Known intolerance to palbociclib or any of its excipients

Additional Criteria for the Palbociclib Combination (Arm D):

1. Prior therapy with a CDK4/6i in the metastatic setting.
2. Known intolerance to palbociclib or any of its excipients.

Additional Criteria for the Abemaciclib Combination (Arm D):

1. Prior therapy with any CDK4/6i.
2. Known intolerance to abemaciclib or any of its excipients.

Additional Criteria for Ribociclib Combination (Arm D):

1. Prior therapy with a CDK4/6i in the advanced or metastatic setting.
2. Known intolerance to ribociclib or any of its excipients.
3. QTcF values ≥450 msec.
4. Participants who already have or who are at significant risk of developing QTc prolongation, including participants with:

   * Long QT syndrome
   * Uncontrolled or significant cardiac disease including recent (6 months) myocardial infarction, congestive heart failure, unstable angina, and brady-arrhythmias
   * Electrolyte abnormalities (K+, Ca++, Phos, Mg++) ≥Grade 1
5. Participant is currently receiving or received drugs known to prolong QT interval within 14 days or 5 half-lives, whichever is shorter, before the first dose of trial therapy.

Additional Criteria for Capivasertib Combination (Phase 1b and Arm E): Recruitment in this combination will occur only in countries where capivasertib is locally approved and available.

1. Prior treatment with any of the following: AKT, PI3K and mammalian target of rapamycin inhibitors and, for Arm E, fulvestrant.
2. Known intolerance to capivasertib or any of its excipients.
3. QTcF values ≥470 msec or factors that increase the risk of corrected QT interval (QTc) prolongation or risk of arrhythmic events such as heart failure, hypokalemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age, or any concomitant medication known to prolong the QT interval.
4. Clinically significant abnormalities of glucose metabolism as defined by any of the following: Participants with diabetes mellitus type 1; participants with diabetes mellitus type 2 requiring insulin treatment or participants with HbA1c level of >8.0% (63.9 mmol/mol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2026-12-27 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with DLTs Observed During the First Cycle | 28 days
  Number of dose-limiting toxicities during the first cycle
Progression-free Survival | 6 months
  The time from the date of the first dose to the date of the first radiological documentation of disease progression or death, whichever comes first.

SECONDARY OUTCOMES:
Standard Pharmacokinetics (PK) Parameters Including AUC0-tau, Cmax, Tmax, and Ctrough | 36 months
  The plasma PK of elacestrant and each of the combination drugs
Overall Response Rate | 36 months
  Proportion of participants who achieve a best overall response of confirmed partial response (PR) or complete response (CR)
Duration of Response | 36 months
  Time from the date of the first documented CR/PR until the first radiological documentation of disease progression or death
Clinical Benefit Rate | 36 months
  Proportion of participants who have the best overall response with a complete response, partial response or stable disease
Progression-free Survival Rate | 36 months
  Time from the date of the first dose to the date of the first radiological documentation of disease progression or death, whichever comes first
Overall Survival | 36 months
  Time from the date of the first dose to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (118):
- United States (45):
  - Dothan Hematology and Oncology, Dothan, Alabama
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - OPN Healthcare (Arcadia Location), Arcadia, California
  - City of Hope National Medical Center, Duarte, California
  - Glendale Adventist, Glendale, California
  - OPN Healthcare (Los Alamitos Location), Los Alamitos, California
  - Cedars Sinai, Los Angeles, California
  - UCLA UCLA Hem/Onc - Clinical Research Unit, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - TOI Clinical Research, Whittier, California
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Yale School Of Medicine - Smilow Cancer Hospital - Breast Center, New Haven, Connecticut
  - George Washington Cancer Center, Washington D.C., District of Columbia
  - Advent Health (Florida Hospital) - Altamonte Springs, Altamonte Springs, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ocala Oncology, Ocala, Florida
  - Northside Hospital Atlanta Cancer Care, Cumming, Georgia
  - Northwestern Feinberg Scholl of Medicine Prentice Women's Hospital, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - MD Alliance for Multispecialty Research, LLC, Merriam, Kansas
  - New England Cancer Specialists, Scarborough, Maine
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Astera Cancer Care, East Brunswick, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Cooperman Barnabas Medical Center, New Brunswick, New Jersey
  - NYU Langone Health, New York, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - W&IH of RI Breast Health Center of Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center Texas, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Cancer Care Northwest, Spokane Valley, Washington
  - Northwest Medical Specialties (Nwms) - Puyallup - Medical Oncology (Rainier Hematology-Oncology)/Exigent Research Network; LLC, Tacoma, Washington
  - University of WI - Carbone Cancer Center (Phase II only), Madison, Wisconsin
- Argentina (4):
  - Centro Medico Austral, Buenos Aires
  - Hospital Britanico De Buenos Aires, Buenos Aires
  - Cemaic - Centro De Especialidades Medicas Ambulatorias E Investigacion Clinica, Córdoba
  - Centro Oncologico Riojano Integral (Cori), La Rioja
- Macquarie University, Sydney, Australia
- Belgium (4):
  - Institut Jules Bordet, Anderlecht
  - Grand Hôpital de Charleroi - Site Notre Dame, Charleroi
  - Universitaire Ziekenhuizen (Uz) Leuven - Campus Gasthuisberg - Multidisciplinair Borstcentrum (Multidisciplinary Breast Center) (Mbc), Leuven
  - Algemeen Ziekenhuis Nikolaas; VITAZ; Oncologie Klinisch Studiecentrum, Sint-Niklaas
- Brazil (5):
  - ACCG - Hospital Araujo Jorge, Goiânia
  - Clinica Neoplasias Litoral, Itajaí
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Centro Gaucho Integrado de Oncologia; Hematologia; Ensino e Pesquisa - Hospital Mae de Deus/AESC, Porto Alegre
  - Hospital Sirio-Libanes (HSL) - Centro De Oncologia - Sao Paulo, São Paulo
- Czechia (2):
  - Nemocnice Horovice Hospital, Hořovice
  - Fakultni Nemocnice Olomouc, Olomouc
- France (5):
  - Centre Hospitalier Lyon SUD- HCL, Lyon
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Centre de Cancérologie du Grand Montpellier, Rouen
  - Centre Hospitalier Universitaire (Chu) De Toulouse - Institut Universitaire Du Cancer De Toulouse-Oncopole (Iuct-Oncopole) (Institut Claudius Regaud), Toulouse
  - Institut Gustave-Roussy-Umr 981, Villejuif
- Germany (8):
  - Universitaetsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Technischen Universitaet Muenchen (TUM), Klinikum Rechts der Isar, Munich, Bavaria
  - Universitatskinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Marienhospital Bottrop, Bottrop
  - Universitatskinikum Carl Gustav Carus Dresden, Dresden
  - Kliniken Essen-Mitte (KEM), Essen
  - Gesundheit Nordhessen Klinikum Kassel, Kassel
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (2):
  - Semmelweis Egyetem Klinikai Kozpont - Onkologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
- Israel (5):
  - Samson Assuta Ashdod University Hospital - The Institute of Oncology, Ashdod
  - Rambam Heath, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Davidoff Rabin Medical Center, Petah Tikva
  - Sheba Medical Center; Center Israel, Ramat Gan
- Italy (6):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera "Istituti Ospitalieri" Di Cremona, Cremona
  - Istituto Europeo di Oncologia (IEO), Milan
  - Istituto Nazionale Tumori "Fondazione PASCALE", Napoli
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Ospedale Infermi di Rimini - Azienda Unita Sanitaria Locale Della Romagna, Rimini
- Centre Hospitalier De L'Ardenne, Libramont, Luxembourg
- Poland (4):
  - Klinika Onkologii; Wojskowy Instytut Medyczny - Państwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Przychodnia Lekarska "Komed" Roman Karaszewski, Konin
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Med-Polonia Sp. Z o.o., Poznan
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (13):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - IOB Madrd Institute of Oncology Hospital Beata Maria Ana de Jesus, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - NEXT Madrid, Pozuelo de Alarcón
  - Fundacion Instituto Valeciano De Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Arnau De Vilanova, Valencia
- Turkey (Türkiye) (2):
  - Abdurrahman Yurtaslan Oncology Hospital, Ankara
  - Ankara Bilkent City Hospital, Bilkent Campus, Universiteler Mh. (old: Ankara Yildirim Beyazit Universitesi), Ankara
- United Kingdom (5):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Liverpool Hospital, Liverpool
  - North Middlesex University Hospital, London
  - Sarah Cannon Research Institute UK; Ltd, London
  - University College London Hospitals NHS Foundation Trust; The London Clinic - Main Hospital, London